CLINICAL TRIAL: NCT06604377
Title: Model of Predicting Biochemical Recurrence After Radical Prostate Cancer Based on Pre-treatment PSMA PET / MR Image Features
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Head of Otolaryngology, Ruijin Hospital
Other Study IDs: RuijinH 2024-244
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: PET/MR; Prostate cancer; Biochemical recurrence; Multicenter
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Shanghai East Hospital, Tongji University School of Medicine: Patients diagnosed with prostate cancer undergoing PSMA PET/MR examination prior to surgery.
  Interventions: Other: Observe

INTERVENTIONS:
Other: Observe — Ruijin

SUMMARY:
The purpose of this study is to investigate the predictive value of preoperative 18F-PSMA-1007 PET/MR in the predictive effect of biological recurrence (BCR) after radical prostatectomy (RP) for localized prostate cancer (PCa).

DETAILED DESCRIPTION:
Construct a predictive model for biochemical recurrence (BCR) in patients after radical prostatectomy using imaging parameters from preoperative 18F-PSMA-1007 PET/MRI, and compare the predictive performance of this model with existing clinical models. Data from three centers will be collected, with datasets from two centers used as the training set for the selection of predictive factors and model construction, while the dataset from the remaining center will serve as the validation set to assess the predictive performance of the model for BCR after prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically confirmed prostate cancer without other types of malignancy -

Exclusion Criteria:

1.Surgery or endocrine therapy is performed prior to the examination

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Patients diagnosed with prostate cancer undergoing PSMA PET/MR examination prior to surgery
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
18F-PSMA-1007 PET/MR image parameters | Before surgery

SECONDARY OUTCOMES:
Biochemical recurrence-free survival time | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No